CLINICAL TRIAL: NCT03908242
Title: Randomized, Double-blind, Placebo-controlled, Continuous Dosing, Single-center, Evaluation of Safety, Tolerability, and Pharmacokinetic Properties of Salvianolic Acid A Tablets in Healthy Volunteers
Brief Title: Phase I Study of Continuous Administration of Salvianolic Acid A Tablet
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Cui Yimin, Director of Pharmacy, M.D. and Ph.D., Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAA003
Record Dates: First submitted 2019-04-06; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — salvianolic acid A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salvianolic Acid A (Experimental): 2 anticipated doses are 90 mg and 180 mg.
  Interventions: Drug: salvianolic acid A
- Placebo Oral Tablet (Placebo Comparator): Placebo tablets containing no salvianolic acid A will be given to healthy subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: salvianolic acid A — salvianolic acid A/Placebo 90 mg bid; salvianolic acid A/Placebo 180 mg qd
  Arms: Salvianolic Acid A
Drug: Placebo — salvianolic acid A/Placebo 90 mg bid; salvianolic acid A/Placebo 180 mg qd
  Arms: Placebo Oral Tablet

SUMMARY:
Salvianolic acid A has a variety of pharmacological effects, such as: anti-oxidation, scavenging oxygen free radicals, anti-fibrosis, anti-myocardial ischemia, anti-coagulation, anti-thrombosis, anti-tumor, etc. Professor Du Guanhua, at Institue of Materia Medica, Chinese Academy of Medical Sciences, first discovered that salvianolic acid A can alleviate diabetic complications and improve patients' quality of life. With the support of major national science and technology projects, the preclinical research work of salvianolic acid A was completed, and the application was approved by the State Food and Drug Administration (Clinical Approval No.: 2016L06293).The purpose of this study is to assess the safety,tolerability, and pharmacokinetics (PK) of an extended dosing regimen ofsalvianolic acid A: open label, continuous subcutaneous infusion for 7 days were tested as ascending doses of salvianolic acid A from 90mg up to 180 mg.

DETAILED DESCRIPTION:
This was a Phase I repeated incremental doses study in healthy volunteers. A total of 24 subjects was planned to be enrolled. This was performed according to a double blind, randomized, placebo controlled design and included two sequential dose groups of repeat doses. Each group enrolled 12 subjects on salvianolic acid A or placebo (ratio 9 experimental: 3 placebo) and received salvianolic acid A or placebo twice daily (90mg) or daily (180mg) for 7 days, and follow-up to 3 or 4 days.

ELIGIBILITY:
Inclusion Criteria:

* 1) Gender: male or female, healthy volunteers; 2) Age: 18~45 years old; 3) Weight: Male subjects need to weigh ≥ 50kg, female subjects should have ≥ 45kg, body mass index [BMI = weight (kg) / height 2 (m2)] in the range of 19 ~ 25 kg / m2; 4) Subjects must give informed consent to the trial prior to the trial and voluntarily sign a written informed consent form; 5) The subject is able to communicate well with the investigator and is able to complete the trial in accordance with the protocol.

Exclusion Criteria:

* (1) Hepatitis B surface antigen, hepatitis C virus, human immunodeficiency virus and syphilis positive; (2) alcoholics; (3) subjects who took any drug or long-term use of drugs within 2 weeks before screening (4) Blood donors within 3 months prior to the trial; (5) participated in any drug clinical trial within 3 months prior to screening; (6) had a clear history of allergic disease; (7) had central nervous system, cardiovascular Systematic, kidney, liver, digestive tract, lung disease, metabolic and skeletal muscle system with a clear history or other significant disease; (8) pregnant, lactating women; (9) other factors not suitable for participation in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-04-08 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events | 10 or 11 days
Percentage of participants with change from baseline in vital signs | 10 or 11 days
  Heart rate, Blood Pressure，auxillary temperature
Change from baseline in electrocardiograms (ECGs) | 10 or 11 days
  PR interval, QT interval, QTc interval, QTcF, and rhythm abnormalities
Percentage of participants with change from baseline in clinical laboratory parameters | 10 or 11 days
  blood routine, urine routine, biochemical parameters of blood and urine，coagulation tests
Plasma concentrations of salvianolic acid A | 8 days
  To investigate the pharmacokinetics (PK) profile of multiple ascending doses of salvianolic acid A

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, Ph.D, Principal Investigator — Peking University First Hospital
Locations (1):
- Xiaocong Pang, Beijing, China

IPD SHARING:
Plan to Share IPD: No